CLINICAL TRIAL: NCT05444920
Title: The Italian Transthyretin Amyloidosis Web-Network (ITA-WebNet)
Brief Title: The Italian Transthyretin Amyloidosis Web-Network
Acronym: ITA-WebNet
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Paolo Milani, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: AC-019-IT
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: ATTR Amyloidosis
Keywords: amyloidosis; systemic amyloidosis
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims, by generating a large registry of patients with ATTR amyloidosis, including data at diagnosis and during follow up, to describe the natural history of ATTR amyloidosis in a real-world setting and to define and validate prognostic models, response criteria applicable at any point of the disease. The registry will also be used for data sharing and to allow the possibility of a close collaboration amongst the amyloidosis experts of the ARTC and all the physicians around the Country involved in the diagnosis and management of systemic amyloidosis. Thanks to the online registry, the diagnostic facility of the ARTC will be made available to requesting physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected diagnosis of systemic and localized amyloidosis;
2. age .18 years;
3. ability to understand and willingness to sign an informed consent (patients who already sign informed consent for clinical data to be used in retrospective analyses will be accepted);
4. planned (or ongoing) follow-up at participating center.

Exclusion Criteria:

1. Diagnosis of light chain (AL) amyloidosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be entered the database pending on expressing an informed consent of the use of their data for research purposes. Data of deceased patients will be used only if they have expressed their consent to the use of their clinical data
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Establishing an online tool for data-sharing, available for health care providers | 5 years
  Different data (types type of organ involvement, biomarkers of organ damage, date of onset of symptoms, date of diagnosis, type of treatment (if any)) will be shared between the health-care professionals and the panel of experts.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No